CLINICAL TRIAL: NCT06289634
Title: The Influence of Man-made and Natural Sounds on Stress, Anxiety, and Mood
Brief Title: The Influence of Sound on Stress, Anxiety, and Mood
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medgar Evers College, The City University of New York (Other)
Responsible Party: Principal Investigator, Sumeyra Tosun, Assistant Professor, Medgar Evers College, The City University of New York
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pending
Record Dates: First submitted 2024-02-22; First posted 2024-03-04 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-02

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Man-made sounds (Experimental): Participants who listen to man-made sounds (music)
  Interventions: Behavioral: Man-made sounds
- Natural sounds (Experimental): Participants who listen to natural sounds (e.g., ocean, birds, rain)
  Interventions: Behavioral: Natural sounds

INTERVENTIONS:
Behavioral: Man-made sounds — Participants will be asked to listen to the assigned sounds (relaxing music) for 30 minutes a day for 15 days.
  Arms: Man-made sounds
Behavioral: Natural sounds — Participants will be asked to listen to the assigned sounds (birds, ocean, wind) for 30 minutes a day for 15 days.
  Arms: Natural sounds

SUMMARY:
Multiple studies have highlighted music's ability to evoke diverse emotional states. Past research reveals that factors like musical elements, and the environment impact how people respond emotionally to music. For instance, faster tempos tend to heighten arousal, while minor key compositions evoke more arousal compared to major key compositions. In efforts to induce specific emotions post-stress, the research found that both pleasant and sad music aided stress recovery. Similarly, other researchers noted that positively rated music was more effective in reducing stress than negatively rated music, especially low arousal compositions over high arousal ones. Several studies focused on applying music to reduce stress and anxiety. In addition to man-made musical tones, the positive impact of natural surroundings on emotional state has been widely explored. A psycho-evolutionary viewpoint was offered, suggesting that humans have evolved in natural settings, making us inherently attuned to them physically and psychologically. A non-threatening natural environment, rich in aesthetically pleasing elements like visible escape routes, greenery, and water, tends to reduce stress and generate interest. In this study, the researchers are exploring how different sounds-man-made instrumental music versus natural sounds-affect stress, anxiety, and mood among the students of Medgar Evers College. Using an experimental approach, the researchers will assess pretest stress levels (via the perceived stress scale (PSS), anxiety (generalized anxiety disorder (GAD-7), and mood (four-dimensional mood scale (4DMS) among a sample of students. After randomly dividing them into two groups, each group will listen to one of the designated sounds (man-made music or nature sounds) for 30 minutes daily over 15 days. The researchers will then have them retake the stress, anxiety, and mood scales for post-test comparison. Statistical analysis (mixed ANOVA) will help to compare scores within and between groups. Ultimately, this study aims to determine the influence of tonal input on stress and anxiety levels among students, crucial given the significant stress they often experience.

DETAILED DESCRIPTION:
Numerous studies have highlighted music's capacity to elicit a wide range of emotions. Previous research suggests that various factors, including musical elements and environmental context, influence people's emotional responses to music. For instance, quicker tempos generally heighten arousal, while compositions in minor keys tend to evoke more arousal compared to major key compositions. In post-stress emotion induction attempts, it was discovered that both pleasant and sad music aided in stress recovery. Similarly, it was observed that positively rated music was more effective in reducing stress, especially compositions with lower arousal compared to those with higher arousal. Several studies have explored the use of music to reduce stress and anxiety.

Moreover, the positive impact of natural surroundings on well-being has been extensively investigated. A psycho-evolutionary perspective was proposed, suggesting that humans have evolved in natural settings, making us inherently attuned to them both physically and psychologically. A non-threatening natural environment, featuring aesthetically pleasing elements like visible escape routes, greenery, and water, tends to decrease stress levels and generate interest.

The study focuses on exploring how different sounds-man-made instrumental music versus natural sounds-affect stress, anxiety, and mood among students at Medgar Evers College.

The research aims to address the following questions:

* Can man-made instrumental relaxing music reduce stress and anxiety levels?
* Does man-made instrumental relaxing music induce a positive change in mood?
* Can relaxing nature sounds reduce stress and anxiety levels?
* Does relaxing nature sounds induce a positive change in mood?
* Is one of the two sound samples more effective than the other?

Ultimately, this study aims to identify the most effective method for reducing stress and anxiety among students, which is particularly important considering the significant stress levels they often encounter.

The findings will be presented at national or international psychology conventions.

ELIGIBILITY:
Inclusion Criteria:

* Being a student at Medgar Evers College, CUNY
* Being 18 years old or older

Exclusion Criteria:

* Having hearing problems

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2024-04 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Stress | 15 days
  Measured by Perceived Stress Scale (PSS). Individual scores on the PSS can range from 0 to 40 with higher scores indicating higher perceived stress.
Anxiety | 15 days
  Measured by General Anxiety Disorder Scale (GAD-7). The outcome of the questionnaire is reported as a score between 0 and 21 with 0 indicating no anxiety and 21 indicating the highest level of anxiety.
Mood | 15 days
  Measured by Four Dimension Mood Scale (4DMS), It is designed to measure positive energy (4 items-minimum score is 4 and maximum score is 20), tiredness (5 items, minimum score is 5 and maximum score is 25), negative activation (6 items-minimum score is 6 and maximum score is 30), and relaxation (5 items-minimum score is 5 and maximum score is 25). Higher scores indicate greater appearance of the corresponding mood.

CONTACTS AND LOCATIONS:
Overall Officials: Sumeyra Tosun, Principal Investigator — Medgar Evers College

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sokhadze EM. Effects of music on the recovery of autonomic and electrocortical activity after stress induced by aversive visual stimuli. Appl Psychophysiol Biofeedback. 2007 Mar;32(1):31-50. doi: 10.1007/s10484-007-9033-y. PMID 17333313
- [Background] van der Zwaag MD, Dijksterhuis C, de Waard D, Mulder BL, Westerink JH, Brookhuis KA. The influence of music on mood and performance while driving. Ergonomics. 2012;55(1):12-22. doi: 10.1080/00140139.2011.638403. PMID 22176481
- [Background] Wang J, Qiu X, Kulkarni A, Hauer-Jensen M. Calcitonin gene-related peptide and substance P regulate the intestinal radiation response. Clin Cancer Res. 2006 Jul 1;12(13):4112-8. doi: 10.1158/1078-0432.CCR-06-0592. PMID 16818712
- [Background] Ulrich RS. Effects of interior design on wellness: theory and recent scientific research. J Health Care Inter Des. 1991;3:97-109. PMID 10123973